CLINICAL TRIAL: NCT00753740
Title: A Phase II Multi-Center Randomized, Double-Blind, Placebo-Controlled Study of Maintenance IT-101 in Platinum Sensitive Ovarian Cancer Patients Who Received 4-6 Cycles of a 2nd Line Platinum-Based Regimen Without Disease Progression.
Brief Title: Efficacy Study of Maintenance IT-101 Therapy for Ovarian Cancer Patients.
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor trial recruitment
Sponsor: NewLink Genetics Corporation (Industry)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OVAR0801; NCT01565421 (obsolete NCT alias)
Record Dates: First submitted 2008-09-12; First posted 2008-09-16 (Estimated); Last update posted 2020-06-12 (Actual); Status verified 2020-06

CONDITIONS: Cancer; Ovarian Cancer; Solid Tumor
Keywords: Cancer; Neoplasms; Solid Tumor; Ovarian Cancer; Solid Malignancies
MeSH Terms: conditions — Neoplasms; Ovarian Neoplasms | interventions — IT-101; Glucose

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 12mg/m2/dose (Experimental): 12mg per meter squared per dose
  Interventions: Drug: IT-101 (12mg/m2/dose)
- 15mg/m2/dose (Experimental): 15mg per meter squared per dose
  Interventions: Drug: IT-101 (15mg/m2/dose)
- Placebo (Placebo Comparator): 5% dextrose infusion (placebo)
  Interventions: Drug: 5% Dextrose (Placebo)

INTERVENTIONS:
Drug: IT-101 (12mg/m2/dose) — Patients who satisfy the inclusion/exclusion criteria will receive a blinded infusion of IT-101 (12mg/m2/dose) every other week until disease progression.
  Arms: 12mg/m2/dose
Drug: IT-101 (15mg/m2/dose) — Patients who satisfy the inclusion/exclusion criteria will receive an infusion of IT-101 (15mg/m2) every other week until disease progression.
  Arms: 15mg/m2/dose
Drug: 5% Dextrose (Placebo) — Patients who satisfy the inclusion/exclusion criteria will receive an infusion of placebo every other week until disease progression.
  Arms: Placebo

SUMMARY:
This study will assess the effect of IT-101 on delaying cancer progression in patients with platinum sensitive ovarian cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Women between the age of 18 and 78, inclusive;
* Evidence of platinum-sensitive ovarian cancer following the patient's primary treatment(>= 6 months);
* Received a 2nd line platinum-based chemotherapy regimen (4-6 cycles) without evidence of progression;
* May have measurable or unmeasurable disease;
* Eastern Cooperative Oncology Group (ECOG) 0 or 1;
* Ability to understand and the willingness to sign a written informed consent document.

Key Exclusion Criteria:

* Women who are pregnant or lactating;
* Prior treatment with a topoisomerase inhibitor;
* Patients with unacceptable organ and/or hematologic reserve at screening;
* Urine protein of > 500 mg/day or active nephropathy;
* Electrocardiogram (ECG) with evidence of clinically significant conduction abnormalities or active ischemia as determined by the investigator;
* History of pancreatitis within the last 12 months;
* Patients treated with previous high dose chemotherapy or stem cell transplant within the last 5 years;
* Use of any investigational agents within 4 weeks of study enrollment;
* Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, psychiatric illness or other co-morbidity that presents a risk to the patient as determined by the investigator.

Ages: 18 Years to 78 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-10 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
To Compare the proportion of patients without evidence of disease progression at 30 weeks following randomization between IT-101 at 12 mg/m2/dose or 15 mg/m2/dose to a placebo infusion treatment administered every other week. | 30 weeks

SECONDARY OUTCOMES:
Comparison of adverse drug experiences between each treatment | 30 weeks
Compare the frequency of drug-related toxicities between each treatment arm | 30 weeks
Compare Quality of Life (QOL, patient-reported) measures (FACT-O, FOSI) between treatment arms. | 30 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S Berek, MD, MMS, Principal Investigator — Professor and Chair, Department of Obstetrics and Gynecology Stanford University School of Medicine Stanford Cancer Center; Franco Muggia, MD, Principal Investigator — Anne Murnick Cogan and David H. Cogan Professor of Oncology, Director of the Division of Medical Oncology at NYU Medical Center, and Associate Director for Clinical Research
Locations (7):
- United States (7):
  - Decatur Memorial Hospital, Clinical Research Department/ Cancer Care Specialists of Illinois, Decatur, Illinois
  - University of Minnesota Medical Center, Minneapolis, Minnesota
  - Schwartz Gynecologic Onclology, PLLC, Brightwaters, New York
  - Gabrail Cancer Center, Canton, Ohio
  - Chattanooga GYN Oncology, Chattanooga, Tennessee
  - The Methodist Hospital, Houston, Texas
  - Riverside Gynecology & Oncology, Newport News, Virginia

REFERENCES:
- [Background] Schluep T, Hwang J, Cheng J, Heidel JD, Bartlett DW, Hollister B, Davis ME. Preclinical efficacy of the camptothecin-polymer conjugate IT-101 in multiple cancer models. Clin Cancer Res. 2006 Mar 1;12(5):1606-14. doi: 10.1158/1078-0432.CCR-05-1566. PMID 16533788
- [Background] Schluep T, Cheng J, Khin KT, Davis ME. Pharmacokinetics and biodistribution of the camptothecin-polymer conjugate IT-101 in rats and tumor-bearing mice. Cancer Chemother Pharmacol. 2006 May;57(5):654-62. doi: 10.1007/s00280-005-0091-7. Epub 2005 Aug 26. PMID 16133526
- [Background] Cheng J, Khin KT, Davis ME. Antitumor activity of beta-cyclodextrin polymer-camptothecin conjugates. Mol Pharm. 2004 May-Jun;1(3):183-93. doi: 10.1021/mp049966y. PMID 15981921
- See also: Calando Pharmaceuticals Website — http://www.calandopharma.com/